CLINICAL TRIAL: NCT06177197
Title: Bronchiolitis Clearance Airways With Seaserum : a Doubled Blind Randomized Study
Brief Title: Bronchiolitis Clearance Airways With Seaserum
Acronym: B-CLASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29BRC23.0193
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Bronchiolitis Acute
Keywords: Infant; Nasopharyngeal decongestion; Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Abortion, Induced

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, controlled, randomized in two parallel arms, double label blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: neither the patient, the parents nor the investigating physician are aware of the product allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiomer (Experimental): It is a sterile, isotonic seawater-based solution, with a concentration equivalent to 9 g/L sodium chloride. This solution is packaged in 5 mL single-dose units.
  It is a Class IIa medical device manufactured by Laboratoire de la mer, and is CE marked.
  Electrodialyzed seawater solution is administered via the nasal passage, in line with current recommendations. Dosage varies according to age, and the pressure exerted on the unit dose enables the product to be administered into the nostril.
  Interventions: Device: Physiomer
- Saline solution (Active Comparator): It is a sterile, isotonic seawater-based solution, with a concentration egal to 0,9 g/L sodium chloride. This solution is packaged in 5 mL single-dose units.
  It is a Class IIa medical device manufactured by GiLBERT, and is CE marked. The saline solution is administered via the nasal passage, in line with current recommendations. Dosage varies according to age, and the pressure exerted on the unit dose enables the product to be administered into the nostril.
  Interventions: Device: Saline solution

INTERVENTIONS:
Device: Physiomer — Infants randomized to the experimental group will be given an electrolyzed seawater solution by their parents for up to 10 days. Dosage is adapted according to the child's age and discomfort:
  * Infant < 6 months: half a dose to a single dose administered per nostril 8 times a day.
  * Infant > 6 months: one single dose administered per nostril 6 times a day.
  Other Names: Electrodilysed seawater solution
  Arms: Physiomer
Device: Saline solution — Infants randomized to the control group will be given a saline solution by their parents for up to 10 days. Dosage is adapted according to the child's age and discomfort:
  * Infant < 6 months: half a dose to a single dose administered per nostril 8 times a day.
  * Infant > 6 months: one single dose administered per nostril 6 times a day.
  Arms: Saline solution

SUMMARY:
The objective of this study is to show that the use of electrodialyzed seawater reduces the duration (in days) of symptoms in acute infant bronchiolitis compared with the use of saline solution in infants aged 1 month to less than one year.

B-CLASS study is a multicenter, prospective, controlled, randomized, double label blind.

DETAILED DESCRIPTION:
This is a multicenter, prospective, controlled, randomized in 2 parrallel arms, double blind study. The Infants will be included after written informed consent will be obtained from the patients' parents or legally authorized representatives. Patients will be randomized either in the experimental group (electrodialyzed seawater) or in the control group (saline solution).

Patients' parents will be call by phone at day 1, day 3, day 6, day 10 and day 21 after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged more than 1 month and less than 1 year
* First episode of acute bronchiolitis
* Emergency consultation
* Existence of nasal obstruction
* Onset of symptoms < 48 hours before emergency consultation
* Outpatient care after emergency consultation
* Mild to moderate bronchiolitis according to the "Haute Autorité de Santé 2019" criteria:

Respiratory rate over 1 minute >30/minutes and <60/minute ; Heart rate >80/minutes and <180/minutes; Absence of respiratory pauses; Absence of superficial breathing; Absence of signs of intense respiratory struggle: involvement of the lower intercostal accessory muscles, sternocleidomastoid muscles, thoracoabdominal swinging, or flapping of the wings of the nose; Feeding >50% of the usual quantity over 3 consecutive doses; SpO2 > 92% during sleep ; >94% when awake; >2 months corrected age

* Parental consent
* Affiliate to a social security system

Exclusion Criteria:

* Hospitalization (excluding short stay unit) after emergency consultation
* Oxygen therapy
* History of prematurity (birth <36 weeks of amenorrhea)
* History of invasive ventilation in the neonatal period
* History of chronic pulmonary or cardiac pathology
* History of immune deficiency
* History of polyhandicap or neuromuscular pathology
* History of malformative Ear Nose and Throat pathology affecting the upper airways
* Impossibility of ensuring the follow-up made necessary by participation in this study

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 458 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Duration of resolution of illness (ROI) | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  It is the time it takes for the child to return to baseline according to the person administering the care.
  ROI is defined by ordinal scale from 0 to 4 on which parents globally rate symptoms according to the following categories: (1) worsened, (2) same, (3) improved, (4) resolved. The duration of ROI is the time it takes to obtain a score of 4.

SECONDARY OUTCOMES:
An again medical consultation | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Have you seen a doctor today for bronchiolitis?" YES/NO
Hospitalization | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Is your child in hospital?" YES/NO. If yes, the length of hospital stay in hours will be collected.
Time to improvement of cough in days | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "How is the cough today?", with four possible answers (1) worsened, (2) same, (3) improved, (4) resolved.
Time to improvement of nasal congestion in days | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "How are colds today??", with four possible answers (1) worsened, (2) same, (3) improved, (4) resolved.
Length with nasopharyngeal decongestion in days | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "How many nasopharyngeal decongestion did you make today?". The duration of nasopharyngeal decongestion is the time it takes to obtain a score of 0.
Number of nasopharyngeal decongestion by day | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "How many nasopharyngeal decongestion did you make today?".
Length of dietary resumption greater than 2/3 of usual intake. | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "How does your child eat today?". Two responses are possible : More than two-thirds, less than two-thirds.
  The duration of dietary resumption greater than 2/3 of usual intake is the number of days until the response is "More than half".
Antibiotic use | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Is your child taking antibiotics?". YES/NO
Length of community eviction en days | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Did your child have to be looked after today?". YES/NO. The duration of community eviction is the time to the child doesn't need to be looked after anymore.
Length of parental absence from work (in days) | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Did you have to miss work today?". YES/NO. The duration of parental absence is the number of day until that parent returns to work.
Occurrence of secondary events: epistaxis, vomiting, malaise, apnea | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Have you noticed any side effects from nasopharyngeal decongestion?". YES/NO.
Time to improvement in respiratory discomfort in days | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "Is your child suffering from respiratory problems today?", with four possible answers (1) worsened, (2) same, (3) improved, (4) resolved.
Time to improvement in sleep quality in days | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Parents will be given a notebook to fill in on a daily basis. For this outcome, the following question will be asked: "How do you rate the quality of your child's sleep?", with four possible answers (1) worsened, (2) same, (3) improved, (4) resolved.
Decrease of number of acute middle ear | At day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10
  Number of patients with an acute middle ear

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Brest, University Hospital, Brest
  - Le Mans hospital, Le Mans
  - Lille, University hospital, Lille
  - Saint-Joseph hospital, Marseille
  - Morlaix hospital, Morlaix
  - Nantes, University Hospital, Nantes
  - Rennes, University hospital, Rennes
  - Tours, University hospital, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.